CLINICAL TRIAL: NCT01214928
Title: Oral Cholecalciferol (Vitamin D3) Therapy in Prevalent Hemodialysis Patients: A Randomized Placebo Controlled Pilot Study
Brief Title: Hemodialysis Vitamin D Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Dr. Catherine Clase, Nephrologist, Associate Professor, St. Joseph's Healthcare Hamilton, McMaster University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJH PSI 001
Record Dates: First submitted 2010-08-30; First posted 2010-10-05 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Vitamin D Deficiency; Renal Failure Chronic Requiring Hemodialysis
Keywords: vitamin D; cholecalciferol; hemodialysis; randomized controlled trial; pilot
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Active Comparator): Cholecalciferol 50,000IU po once weekly for 12 continuous weeks.
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): Matching placebo po once weekly for 12 continuous weeks
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — cholecalciferol 50,000 IU po once weekly for 12 weeks
  Other Names: vitamin D3

SUMMARY:
Vitamin D is a prohormone obtained through diet, supplementation, or sun exposure. Once absorbed, this nutritional vitamin D undergoes a two-step reaction in the liver and in the kidney to become the active hormone, calcitriol. Besides the kidney, many other body tissues are capable of local vitamin D activation. This local tissue activity is important for maintenance of health and relies on adequate levels of nutritional vitamin D. Not only are dialysis patients deficient in calcitriol due to kidney failure, but they are also deficiency in nutritional vitamin D. Low levels of vitamin D have been associated with higher rates of death, heart and blood vessel disease, osteoporosis, falls, cancer, and autoimmune diseases. Despite this, there is a lack of randomized controlled trials (RCT) examining the effects of nutritional vitamin D in hemodialysis (HD) patients. The investigators hypothesize that long-term supplementation with nutritional vitamin D in HD patients improves survival and cardiovascular outcomes. Before embarking on a large scale RCT, the investigators propose a small pilot RCT with 20 hemodialysis patients to: i) To determine the effects of cholecalciferol (vitamin D3) in raising blood vitamin D levels; ii) To determine the feasibility and barriers to successful randomization and adherence to treatment protocols, which will inform subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 18 years
2. Participant is on hemodialysis ≥ 3 months

   Exclusion Criteria:
3. Serum calcium >2.75 mmol/L
4. On concurrent vitamin D treatment ≥ 800 IU/day. Includes ergocalciferol, cholecalciferol, calcedidiol, over-the-counter vitamin D. Does not include one-alpha calcidol (One Alfa®) or 1, 25 di-hydroxy-D3 (Rocaltrol® or Calcijex®)
5. Known hypersensitivity or allergy to Vitamin D
6. End stage liver disease
7. Severe untreated malabsorption or resection of large segment of small bowel
8. Lack of informed consent or inability to consent
9. Currently enrolled in a RCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Feasibility objectives for this proof-of-concept study | 1 year
  1. To determine the proportion of consecutive HD patients that are eligible, the proportion of eligible patients that will consent to randomization, and of those randomized, the proportion that will comply with their group assignment.
  2. To determine the treatment effect of oral cholecalciferol compared with placebo in raising serum 25(OH)D and 1,25(OH)2D levels in HD patients.

SECONDARY OUTCOMES:
Six Minute Walk Test | 1 year
  1. To determine the proportion of eligible patients that are able to complete a baseline and end of study 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Karen CY To, MD, FRCPC, Principal Investigator — St. Joseph's Health Care London; Catherine Clase, FRCPC, Principal Investigator — St. Joseph's Health Care London; Azim S Gangji, MD, FRCPC, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada